CLINICAL TRIAL: NCT01292161
Title: Study of Silymarin for Improving Hepatitis C
Brief Title: Effects of Silybum Marianum on Treatment of Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy, Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-15
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2006-09

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Silymarin; Quality of life
MeSH Terms: conditions — Hepatitis C | interventions — Silymarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Silymarin (Other): Silymarin drived from Silybum marianum (milk thistle), a flowering member of the daisy family, may benefit liver function in people infected with the hepatitis C virus.
  Interventions: Drug: Silymarin

INTERVENTIONS:
Drug: Silymarin — Tab 210 mg, 630 mg, daily, six months.

SUMMARY:
The purpose of this study is to determine the effects of silymarin on outcomes of patients with hepatitis C.

DETAILED DESCRIPTION:
Silymarin has been claimed to have a beneficial effect in various types of liver injury, including alcoholic liver disease, drug and toxin induced hepatotoxicity, and acute and chronic viral hepatitis.

ELIGIBILITY:
Inclusion Criteria:

confirmed chronic hepatitis C (HCV Ab (+), HCV RNA (with PCR) (+)) normal or increased liver enzymes (ALT and AST) not using interferon or ribavirin due to patient sensitivity or not consenting.

Exclusion Criteria:

The pregnant patients patients with side effect which confirmed with rechallenge test

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Serum aminotransferases (ALT, AST) | at six months after admission
  The investigators measured serum amino transferases by commercial AST kit,. ALT kits(Bayer Diagnostics,. Tarrytown, NY, USA) at six months after silymarin admission

SECONDARY OUTCOMES:
HCV-RNA | at six months after admission
  The investigators measured serum HCV-RNA by Polymerase Chain Reaction (PCR) at six months after silymarin admission

CONTACTS AND LOCATIONS:
Overall Officials: hamid kalantari, A.Professor, Principal Investigator — Associate Professor,Gasteroentrology department
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran

REFERENCES:
- See also: Isfahan university of medical sciences — http://mui.ac.ir